CLINICAL TRIAL: NCT02233465
Title: Mesh-repair With Inraperitoneal On-lay Mesh (IPOM) for Parastomal Hernia
Brief Title: Treating Parastomal Hernia With a Mesh
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Norrbottens Lans Landsting (Other)
Responsible Party: Principal Investigator, Pia Nasvall, MD, Norrbottens Lans Landsting
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-021M
Record Dates: First submitted 2014-05-12; First posted 2014-09-08 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Parastomal Hernia
Keywords: parastomal; hernia; mesh; parastomal hernia-repair with mesh
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IPOM Mesh-repair parastomal hernia (Experimental): Mesh-repair of para-stomal hernia. Patients with para-stomal hernia requiring surgery are offererd enrollment in the study. Preoperatively a CT-scan of the abdomen and or a 3D ultrasonography of the stoma is performed. All patients in the stydy are operated with IPOM-mesh designed for treatment of parastomal hernia.
  Interventions: Procedure: IPOM Mesh-repair parastomal hernia
- No mesh-repair (No Intervention): Patients not attending the study

INTERVENTIONS:
Procedure: IPOM Mesh-repair parastomal hernia — Safety study for mesh-repair of parastomal hernia
  Other Names: Device: Parastomal hernia patch BARD
  Arms: IPOM Mesh-repair parastomal hernia

SUMMARY:
Parastomal herniation is difficult to treat. Several different treatment has been tested but still none has revealed to be superior. The use of a mesh has been shown to be a promising way of treating. In this study the investigators will evaluate safety and hernia recurrence rate with a mesh tailored to treat parastomal hernias "Parastomal hernia mesh BARD" in patients with parastomal hernia requiring surgery.

DETAILED DESCRIPTION:
Parastomal hernia is a common complication in patients with a stoma and may cause the patient difficulties with stomal dressing and leakage of stomal content, as well as pain and risk for incarceration. The exact hernia incidence is not known, it depends on the definition of whether a bulge is considered a hernia or not, as well as the duration of follow-up. The reported incidence ranges between 0 and 52%. The majority of parastomal hernias develop within a few years after the index operation, but can appear as late as 20 years after surgery.

There is no superior treatment for an existing parastomal hernia. Several methods have been tested and used such as stoma relocation, sutures to narrow the opening in the fascia and abdominal wall and fixation and closure of the lateral space but none has proven to prevent from recurrence of herniation. Mesh repair has been shown to give a lower recurrence rate 0-33%. No technical factor, such as site of stoma formation (through or lateral to rectus abdominis muscle), related to the construction of the stoma was proven to prevent hernia formation.

To find a way to prevent the occurrence of parastomal hernia is an important issue. Today there are reports proposing a mesh in sublay position at the index operation would prevent hernia formation. Although the results are promising these studies are small and they do not meet the issue late complications according to the mesh implant.

The use of intraperitoneal on-lay mesh (IPOM) is widely used to treat incisional hernia. A new mesh (Parastomal hernia mesh BARD) has been tailored to treat parastomal hernia. To evaluate safety and hernia recurrence rate using the BARD-mesh for treating parastomal hernia a prospective multicentre non-randomised study is performed. The aim is to include 50 patients in the study.

Patients with parastomal hernia requiring surgery due to leakage, problems with stoma dressing, bulging, incarceration and other problems related to the hernia will be offered enrollment in the study after informed consent. The preoperative examination include clinical examination, three dimensional ultrasonography (3D) and or computed tomography (CT) of the abdomen.

Surgery at the four hospitals will be performed by experienced colorectal surgeons with a special interest in parastomal hernias. Postoperatively the patients will be allowed to mobilize according to each hospital postoperative routines. Follow-up visits at one month, one year and three year are scheduled. Early complications like infections, ileus, myocardial infarction, pneumonia, urinary infection and thrombosis are evaluated at one-month follow-up by clinical examination. At one and three year follow-up late complications and possible recurrence of parastomal hernias will be searched for. CT will be performed one year postoperatively. At the three year follow-up CT and or 3D will be performed.

Important outcome measures are complications and recurrence of parastomal hernia.

ELIGIBILITY:
Inclusion Criteria:

* Parastomal hernia requiring surgery, over the age of 18

Exclusion Criteria:

* Patient not accepting participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Parastomal recurrence rate | One year and three year

SECONDARY OUTCOMES:
Complications | three months, one year and three year

CONTACTS AND LOCATIONS:
Overall Officials: Pia Näsvall, MD, Principal Investigator — Dep of Surgical and Perioperative Sciences, Umeå University